CLINICAL TRIAL: NCT03853954
Title: Reduction of Anterior Shoulder Dislocation Facilitated by Inhaled Low Dose Methoxyflurane - a Pilot Study
Brief Title: Reduction of Anterior Shoulder Dislocation Facilitated by Inhaled Low Dose Methoxyflurane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CapitalDHACCanada
Record Dates: First submitted 2019-02-22; First posted 2019-02-26 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Shoulder Dislocation
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Intervention Model Description: This prospective open-label pilot study will examine the use of inhaled low dose methoxyflurane to facilitate shoulder reduction in a convenience sample of patients arriving with anterior shoulder dislocations. This study will test the feasibility of studying the addition of this analgesic agent to a reduction technique that classically eschews procedural sedation in order to increase successful reduction rates. Consenting eligible patients will be offered a first attempt at reduction using the method described by Cunningham, supported by self-administered low-dose methoxyflurane analgesia as instructed by the advanced/critical care paramedic. For unsuccessful first attempts, patients will then undergo the current standard of care for shoulder dislocations, which is reduction of the shoulder joint while under procedural sedation and analgesia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Methoxyflurane (Experimental): Dosage form: inhalation Dosage: 3 mL methoxyflurane per inhaler, to be self-administered Frequency: maximum one inhaler (3 mL) per patient Duration: <15 minutes
  Interventions: Device: Methoxyflurane

INTERVENTIONS:
Device: Methoxyflurane — Methoxyflurane (Penthrox) inhaler, 3mL inhalation vapour, liquid
  Other Names: Penthrox

SUMMARY:
This pilot study will test the feasibility of doing a definitive study to ascertain whether reduction of shoulder dislocation can be safely and effectively facilitated by a patient controlled inhalational analgesic, negating the need for potentially dangerous PSA and the use of intravenous therapy. The hypothesis includes that time to reduction and time spent in the emergency department will be reduced.

DETAILED DESCRIPTION:
Anterior shoulder dislocation, in which the head of the humerus (cup) comes out of its position in the glenoid fossa (saucer), to lie anterior and below its proper position, is a common emergency department presentation. Between April 1, 2011 and March 31, 2018, 1654 patients presented to emergency departments in Emergency Departments of the Central Zone of the Nova Scotia Health Authority (Average 236/year). The treatment of dislocated shoulder involves reduction to a normal anatomical position as soon as possible, to manage pain and disability and to minimize the chance of poor long term outcome. Numerous methods exist to effect reduction, most of which are conducted under procedural sedation and analgesia (PSA) that allows the shoulder muscles to relax so that they do not hold the humeral head in a dislocated position. PSA involves the administration of intravenous sedatives and narcotic analgesics. Not only do the medications carry the risk of respiratory depression and hypotension, but their duration of action results in longer emergency department stays and the use of intravenous lines, is invasive and adds patient discomfort and expense to the procedure. An additional risk of PSA in this specific population is that reduction of the dislocation to its normal position, immediately removes the painful stimulus that antagonizes the respiratory depression of the sedative and analgesic agents. This often results in unopposed respiratory depression which might be unrecognized as the 'crisis' appears to be over with the restoration of the shoulder joint. Furthermore, PSA requires specifically trained staff and space; and time taken to arrange PSA prolongs the time during which the humerus is out of position. It has been reported that from the time of arrival in the emergency department with an anterior shoulder dislocation, every 10 min delay in reduction attempt increased the odds of a failed reduction attempt by 19%. In the Charles V. Keating Emergency and Trauma Centre in Halifax, Nova Scotia, PSA is conducted by specially trained advanced care paramedics using standard preparation, monitoring and recovery protocols. In an effort to painlessly reduce shoulder dislocations without PSA, the Cunningham technique has been described, which involves massaging the shoulder muscles in an attempt to get them to relax sufficiently to allow reduction. Although this method does work, and has been associated with decreased need for PSA, it is associated with an increase in the rate of unsuccessful first reduction attempts. After unsuccessful attempts using the Cunningham technique, the fallback is generally to then provide PSA, increasing the time to reduction. Inhaled low-dose methoxyflurane has been used for several decades in Australia as an emergency analgesic for short-term use. Administered via a portable, disposable, single-use hand-held inhaler device administered by the patient for pain relief, it offers a safe and effective non-opioid alternative to morphine. Inhaled methoxyflurane has been shown to be safe, effective, and simple to administer in obstetric patients during childbirth, as well as for patients with bone fractures and joint dislocations, and for dressing changes on burn patients. In 2018, PenthroxTM (methoxyflurane) received marketing authorization from Health Canada for adult patients requiring short-term relief from moderate to severe acute pain associated with trauma or interventional medical procedures. Low dose methoxyflurane adds to the armamentarium of Canadian emergency care providers as an option that is relatively inexpensive, safe and very easy to administer rapidly. As most failures of the Cunningham anterior shoulder reduction method are due to patient discomfort, the investigators hypothesize that inhaled low dose methoxyflurane has the potential to increase first attempt success rates using this method while decreasing the time from arrival to reduction, the need for intravenous therapy or the use of potentially dangerous medications. The Penthrox inhalers will be supplied by Purdue and will be stored in the emergency department in a locked cabinet in a locked box with limited access. It is a self controlled inhaled medication controlled by each inhalation. Each breath a patient takes releases a fraction of the single dose contained in the inhaler.

ELIGIBILITY:
Inclusion Criteria:

* Anterior dislocation not complicated by fracture (pre-reduction x-rays will be done at the discretion of the emergency physician)
* No neurological or vascular injury
* Patients greater than or equal to 18 years of age
* Patients able to understand the nature of the study and give written informed consent
* Patient is able to follow all study requirements and procedures and complete all questionnaires

Exclusion Criteria:

* Previous shoulder surgery on the affected side
* Associated fracture or secondary significant injury
* Previous in-hospital reduction attempt for the current dislocation
* Open wound or infection in the vicinity of the joint
* Uncorrectable altered level of consciousness, to be defined by the attending clinician as a Glasgow-Coma Scale of less than 15, due to any cause, including head injury, drugs, or alcohol
* History of clinically significant renal impairment
* History of liver dysfunction after previous methoxyflurane use or other halogenated anesthetics
* Hypersensitivity to methoxyflurane or other halogenated anesthetics
* Known or genetically susceptible to malignant hyperthermia or a history of severe adverse reactions in either patient or relatives
* Clinically evident hemodynamic instability
* Clinically evident respiratory impairment
* Has received methoxyflurane within the past 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Incidence of first reduction attempt success | Minutes from the beginning of procedure (maximum 15 minutes)
  'First attempt' will be defined as 'That before a decision is made to try a different method of reduction' - i.e. a pause during the attempt to allow further muscle relaxation and analgesia will not imply failure of the first attempt however if no success at the 15-minute mark, the procedure will be aborted and standard PSA will be conducted for further reduction attempts.
Time of arrival to beginning of first reduction attempt | Up to a maximum of 24 hours from emergency department registration
  Documented triage time to time of methoxyflurane administration.

SECONDARY OUTCOMES:
Time to discharge from ED | Up to a maximum of 24 hours from emergency department registration
  Documented triage time to time patient is ready for discharge
Provider satisfaction with the process | Completed within 30 minutes of intervention
  5-Point Likert scale of provider satisfaction with process: 1-poor, 2-fair, 3-good, 4-very good, 5-excellent
Treatment-related adverse events | Up to a maximum of 24 hours from emergency department registration
  Incidence of the following treatment-related adverse effects in the study population: hypotension (SBP <100 mmHg OR <85 mmHg if baseline SBP <100 mmHg), vomiting, somnolence, amnesia, dizziness, headache, cough, other (document), none

CONTACTS AND LOCATIONS:
Overall Officials: Samuel G Campbell, MD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- NSHA, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No